CLINICAL TRIAL: NCT04110015
Title: Assessment of Visual Function in Ophthalmic Disorders Using Virtual Visual Field Analysis
Acronym: proVVF
Status: Terminated | Type: Observational
Why Stopped: New heightened internet security at HHC and VVF device no longer compliant with intranet and internet access at hospital
Sponsor: New York City Health and Hospitals Corporation (Other)
Responsible Party: Principal Investigator, Joyce Mbekeani, Associate Professor of Ophthalmology & Visual Sciences, New York City Health and Hospitals Corporation
Other Study IDs: 2019-10418
Record Dates: First submitted 2019-09-21; First posted 2019-10-01 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Visual Pathway Disorder; Glaucoma; Retinal Disease
MeSH Terms: conditions — Glaucoma; Retinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Neurology patients: Any patients with neurological disorders
  Interventions: Device: virtual visual field
- Glaucoma patients: Any patients with chronic open angle and chronic angle closure glaucoma of all stages
  Interventions: Device: virtual visual field
- Retina patients: Any patients with known retinal conditions
  Interventions: Device: virtual visual field

INTERVENTIONS:
Device: virtual visual field — Patients with identified conditions will be invited to do a virtual visual field test with virtual reality headsets.

SUMMARY:
1. To evaluate the accuracy of virtual visual field (VVF) headsets equipped the standard visual field software in its ability to assess visual function in various retinal, glaucoma and neuro-ophthalmic disorders by comparing retinal fundus and optic nerve images, optical coherence tomography and neuroimages to the VVF produced.
2. To test the null hypothesis that VVF testing compares favorably to the gold standard, Humphrey visual field (HVF) by comparing testing time, mean sensitivity, markers of reliability including false positives and negatives and fixation losses and global indices such as mean deviation and pattern standard deviation.

DETAILED DESCRIPTION:
1. Study Style: Prospective, Controlled Clinical Trial
2. Objectives:

   1. To determine the capacity for a portable head-mounted virtual visual field-testing device, with capacity for remote testing, to accurately analyze visual function in various retina, neuro-ophthalmic and glaucoma disorders.
   2. To compare virtual visual field results with the "gold standard," Humphrey visual fields.
3. Subjects: Consecutive patients already scheduled for visual fields for various retina, glaucoma and neuro-ophthalmic conditions and normal controls.

SETTING AND PROTOCOL FOR HUMAN RESEARCH:

1. Location: Ophthalmology Department, Jacobi Medical Center, Bronx New York.
2. Recruitment: Patients already presenting to the eye clinic or seen on the wards at Jacobi Medical Center will be offered a chance to participate as volunteers. No other active recruitment will be done.
3. Retention and Dropout: Investigators will encourage patients to complete their testing. However, it will be made clear that they can drop out at any time without need to provide a reason. Dropouts will be replaced with other consenting patients.
4. Protocol (Interventions and Timing):

   1. Consecutive patients presenting to the Jacobi eye clinic and wards who are diagnosed with neurologic, glaucoma and retina conditions and already are scheduled to have Humphrey visual field analysis, will be asked if they would like to voluntarily participate in this study.
   2. Interested patients will be have the study explained to them and an informed consent taken by the study resident/technician.
   3. The standard Humphrey visual field (HVF) will be conducted by the technician (5-10 minutes) in the usual manner.
   4. The option of doing the virtual fields immediately, on the same day, will be offered vs returning to conduct the test within 3 months.
   5. The virtual reality headset will be applied and instructions in the patient's preferred language provided through the earpiece of the virtual visual field (VVF). When the patient indicates they wish to proceed, the test will be started by the technician.
   6. The technician is already versed in conducting both versions of the visual field tests.
5. Clinical Analysis: All fields will be stored digitally within each Health Insurance Portability and Accountability Act (HIPAA) compliant device-specific website for later analyses by respective Attendings (glaucoma, retina and neuro-ophthalmology/neurology).
6. Data Collection:

   1. The patients' demographic details, visual field pattern deviation, and global indices (mean deviation, f and pattern standard deviation) and reliability indices (fixation losses, false positives/negatives will be documented in the data collection Excel sheet.
   2. Supporting ancillary tests (optical coherence tomography, retina photography and neuroimaging) will be collected for each patient and reported findings documented. These tests are part of normal standard of care assessment of patients at Jacobi Medical Center.

STUDY POPULATION:

1. Consecutive clinic and ward patients (>18yrs old) with glaucoma, retinal or neurological disorders able to understand, consent and deemed physically able to perform the visual field tests.
2. Power Calculation:

   1. Alpha 0.05
   2. Power 80%
   3. Using the findings of mean deviation (MD) in perception of light from a previous VVF glaucoma study : mean (SD)=-3.78 (7.49) dB units in glaucoma patients and 0.587 (2.588) dB in the controls.
   4. 39 patients and 39 controls in each sub-population (retina, glaucoma and neuro-ophthalmology) will be required to sufficiently power the study. Round numbers of 40 cases and 40 controls for each study to be sufficiently powered.

For all three studies, 120 study cases in total will be tested with clinical conditions and 120 normal cases as normal controls. 240 cases in total will be tested.There will be confounding variables that can be addressed with subgroup analysis or multivariate regression analysis.

INFORMED CONSENT:

1. The informed consent to participate in the study will be taken at the site of testing at Jacobi Medical Center.
2. The informed consent will be taken by one of the study residents or the study technician.

STATISTICAL ANALYSIS: Excel and SAS (Statistical Analysis Software, SAS institute Inc. Cary, North Carolina, USA) software will be used for descriptive assessment and statistical analysis of the data set and generation of graphs.

1. Data will be used to test the hypothesis that the virtual visual field headset is able to accurately detect visual field defects in ophthalmic conditions and develops visual field maps and global indices that compare favorably with the gold standard, Humphrey visual fields.
2. Interim analyses will be conducted for each sub-population (glaucoma, retina, neurology) when they reach the power number ~40.
3. Once all data is de-identified, it will be analyzed using SAS software.
4. Descriptive data will be determined with basic percentages.
5. Aggregate means of global indices of each study group: retina disorders, glaucoma of all stages (1-mild; 2-moderate; 3-severe; 4-indeterminate) and neuro-ophthalmic conditions, will be compared with their control group and VVF compared to HVFusing t-test, Chi-square, Mann-Whitney and Kruskal-Wallis tests.
6. Correlation between the parameters of virtual visual field test and Humphrey visual field including time for test, mean sensitivity (MS, expressed in decibels), fixation loss (FL), false negative (FN), false positive (FP), mean deviation (MD) and pattern standard deviation (PSD) will be assessed using linear regression models that will account for confounding variables such as age, visual acuity and other ocular conditions.
7. Statistical significance will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with retina, glaucoma and neuroophthalmic disorders
* Patients with normal eye exams to act as controls
* Must be able to comprehend instructions and perform visual fields

Exclusion Criteria:

* Patients <18years old
* Patients unable to comprehend visual field instructions or unwilling to participate
* Patients lacking a complete clinical file or lacking a specific diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All consecutive patients (>18yrs old) with glaucoma, retinal or neurological disorders able to understand, consent and deemed physically able to perform the visual field tests.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-08-23 (Actual)

PRIMARY OUTCOMES:
Virtual visual field result | with 3 months
  Gray scale pattern will reveal areas of vision loss or visual depression; this will have a numerical total deviation plot giving numbers in decibels of the points in the visual field of depressed or lost points of vision. Global indices also will be recorded; these give numerical quantification in decibel units of visual field loss. and include: mean deviation - the average of all decreased perception, pattern deviation which highlights localized losses and pattern standard deviation which quantifies the amount of loss and gauges progression. Time take to complete fields and reliability indices will be recorded: fixation losses, false positives, false negatives
Humphrey visual field result | within 3 months
  Gray scale pattern will reveal areas of vision loss or visual depression; this will have a numerical total deviation plot giving numbers in decibels of the points in the visual field of depressed or lost points of vision. Global indices also will be recorded; these give numerical quantification in decibel units of visual field loss. and include: mean deviation - the average of all decreased perception, pattern deviation which highlights localized losses and pattern standard deviation which quantifies the amount of loss and gauges progression.

SECONDARY OUTCOMES:
Comparison of Virtual Visual field (VVF) to Humphrey visual fields (HVF) | At end of study when we have all the data ~ one year
  Comparison of patterns, global indices and reliability indices between VVF and controls and then VVF and HVF.

CONTACTS AND LOCATIONS:
Overall Officials: JOYCE MBEKEANI, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Jacobi Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share data.